CLINICAL TRIAL: NCT01118858
Title: Exogenous and Endogenous Biomarkers of CYP2D6 and CYP3A4 Variability in Pediatrics
Brief Title: Biomarkers of CYP2D6 and CYP3A4 Variability in Pediatrics
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Steve Leeder, Pharm.D; Ph.D., Children's Mercy Hospital Kansas City
Other Study IDs: 1R01HD058556-01A1 (NIH); 5R01HD058556 (NIH)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Drug Metabolism Phenotype
Keywords: CYP2D6; CYP3A4; cytochrome P450; children; pediatrics; dextromethorphan; phenotype; genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or saliva for DNA testing. Blood samples will be obtained for safety labs throughout the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Pediatric patients who have a primary diagnosis of ADHD, combined type, hyperactive impulsive, or inattentive type (ADD).
- Control: Healthy subjects: Age and gender matched subjects who do not meet any of the exclusion criteria

SUMMARY:
Cytochrome P450 2D6 (CYP2D6) is an important enzyme in the body for breaking down many medications that are commonly used in children of various ages. The purpose of this proposal is to investigate the relative roles of development and genetic variation in CYP2D6 activity in school-aged children and adolescents with attention deficit and hyperactivity disorder and health controls using the over-the-counter cough suppressant, dextromethorphan or "DM", a standard probe for determining CYP2D6 phenotype. Embedded in the study design are sub-studies to search for by-products of normal body metabolism that reflect differences in enzyme activity, and a pharmacokinetic study to assess the consequences of CYP2D6 genetic variation on the systemic exposure to medications used by this patient population. Ultimately, the goal of the research is to personalize the use of medications in children by selecting the appropriate dose of the correct medication for individual patients.

DETAILED DESCRIPTION:
This proposal represents a continuation of previous and ongoing longitudinal studies to characterize the relative contribution of pharmacogenetics and ontogeny to variability in CYP2D6 and CYP3A4 activity between birth and adolescence. Specifically, the overall goal of the research program is to test the hypothesis that genetic variability, rather than ontogeny, is the primary source of variability in CYP2D6 and CYP3A4 activity during adolescence. This study will extend our current series of longitudinal phenotyping studies and will be a cross-sectional study in children aged 7-15 years, studied on seven occasions, 6 months apart.

Children will be recruited from Children's Mercy Hospitals and Clinics, The Children's Mercy Hospital Northland Campus, and The Children's Mercy South Campus.

Subjects participating in this study will consist of a total of 220 children and adolescents from 7 to 15 years of age with a gender and ethnic distribution representative of the patient population served by Children's Mercy Hospital (CMH; from a representative 12 month period) as follows: White, 59.6%; African-American, 31.9%; Hispanic, 4.9%; Asian, 0.6%;Native American, 0.1%; Other, 2.9%. The gender distribution is 44.4% female and 55.6% male. An equal number of pediatric patients who meet the DSM-IV criteria for a primary diagnosis of ADHD or ADD (~33%) and age- and sex-matched controls (~67%) will be recruited. The patients represent a population of children who can reasonably expect to be treated with a medication that is primarily dependent upon CYP2D6 for its elimination from the body. An example is atomoxetine, also known as Strattera®. Each patient will be asked to invite a friend to participate in the phenotyping study with them, providing a non-ADHD population as a reference. Additional phenotyping visits will occur every six months (totaling 7 visits). Justification: Assuming a 10% attrition rate for the second visit, the sample size is expected to provide approximately 25 patients and 25 controls (50 subjects total) in each initial 2-year age bin: 7.0 to 9.0 y, 9.1 to 11.0 y, 11.1 to 13.0 y, and 13.1 to 15.0 y.

Subjects will be enrolled via informed permission/assent and will be studied as outpatients utilizing resources provided by the Pediatric Clinical Research Unit located in the Division of Clinical Pharmacology and Medical Toxicology at Children's Mercy Hospital. For the ADHD group, patients being treated with atomoxetine at the time of study enrollment will be allowed to participate. Although in vitro studies indicate that atomoxetine inhibits CYP2D6 activity by ~50%, there does not appear to be any effect in vivo as single dose pharmacokinetics of the CYP2D6 substrate, desipramine, were unaffected by four days of atomoxetine 60 mg b.i.d. Thus, we do not expect any substantial effect on DM biotransformation. Furthermore, if during the six month interval between phenotyping visits ADHD patients are prescribed medications that are known CYP2D6 inhibitors, they will be allowed to continue in the study; the dose and start date of these medications will be recorded and the effect of the inhibitor on CYP2D6 phenotype (urinary metabolite ratio and endogenous biomarker) will be determined. These data points will be excluded from the ontogeny and genotype-phenotype correlation analysis

Pre-study visit. (about 1 hour long) On a screening visit, prospective subjects (and their parents) will be provided with a description of the proposed study. After all their questions have been answered, they will be given a copy of the permission/assent form to review and sign Subjects will then have their medical history and use of medications reviewed, including the use of non-prescription and herbal remedies. All subjects will be given a complete physical examination by a physician, including vital signs (blood pressure, heart rate, breathing rate, temperature, height and weight) and an assessment of pubertal development by Tanner stage. Breast development will be assessed by visual inspection. Pubic hair will be assessed by visual inspection. Testicular volume will be measured by direct comparison to orchidometer beads. Tanner Staging will be assessed by a gender appropriate physician. Blood will be drawn by needle stick for serum chemistries, liver function tests and a hematology panel; a portion will also be retained for DNA testing (approximately 2 teaspoons of blood total). Urine will be collected for a Urinalysis with Micro. Numbing cream may be applied to the site to minimize discomfort. A urine pregnancy test will be performed for females of child bearing age.

The DNA testing, referred to "genotyping" will be conducted by a combination of technologies designed to detect variations from single nucleotide level (including polymorphisms, insertions and deletions), to larger gene deletions, rearrangements, hybrid structures and copy number variations using established methods in the Developmental Pharmacology and Experimental Therapeutics Laboratory. As next-generation sequencing technology becomes established, existing technologies will be replaced by next-generation sequencing for its ability to assess the entire gene region rather than at individual locations.

Study Day 1 (about 5 hours long) Within approximately one week of the pre-study visit, subjects will be admitted to the study unit. The child must refrain from eating 2 hours prior to the scheduled visit. Prior to dosing, the subjects will completely empty their bladders and provide a blank urine sample. Each subject will then be given a single 0.5 mg/kg dose of DM as Robitussin Cough (7.5 mg/5 ml; alcohol-free, fruit punch flavor). All urine produced over the 4-hour study period will be collected. Urine will be retained for analysis of DM and its three metabolites, and for metabolomic analyses. One hour after dosing, the subjects will be provided with a small meal that they will select from the standard hospital menu. A pregnancy test will be performed for females of child bearing age. Subjects will be asked to provide breaths (inspiratory and expiratory) for ten minutes with a handheld indirect calorimeter (ie. MedGen/Body Gem: also known as "GEM") with a clip on their nose. The measurements obtained for resting metabolic rates will occur prior to dosing and 4 hours post dose.

Subjects will be asked how they are feeling during the study and before going home.

Study Day 2-7 (about 5 hours long) The remaining visits will occur every 6 months following Study Day 1; the study sessions will be delayed for 1-2 weeks if the subjects are suffering from flu-like symptoms. The child must refrain from eating 2 hours prior to the scheduled visit. For females, a pregnancy test will be conducted using the pre-dose urine sample prior to DM dosing.

Subjects will then have their medical history and use of medications reviewed, including the use of non-prescription and herbal remedies. Subjects will be given a complete physical examination by a physician, including vital signs (blood pressure, heart rate, breathing rate, temperature, height and weight) and an assessment of pubertal development by Tanner stage. Breast development will be assessed by visual inspection. Pubic hair will be assessed by visual inspection. Testicular volume will be measured by direct comparison to orchidometer beads. Tanner Staging will be assessed by a gender appropriate physician.

Subjects will be admitted to the study unit. Prior to dosing, the subjects will completely empty their bladders and provide a blank urine sample. Each subject will then be given a single 0.5 mg/kg dose of DM as Robitussin Cough (7.5 mg/5 ml; alcohol-free, fruit punch flavor). All urine produced over the 4-hour study period will be collected. Urine will be retained for analysis of DM and its three metabolites, and for metabolomic analyses. One hour after dosing, the subjects will be provided with a small meal that they will select from the standard hospital menu. A pregnancy test will be performed for females of child bearing age. Subjects will be asked to provide breaths (inspiratory and expiratory) for ten minutes with a handheld indirect calorimeter (ie. MedGen/Body Gem: also known as "GEM" with a clip on their nose. The measurements obtained for resting metabolic rates will occur prior to dosing. Subjects will be asked how they are feeling during the study and before going home.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 7 and 15 years of age.

Exclusion Criteria:

* Inability to have blood drawn for the screening lab tests
* Current therapy with medications known to inhibit CYP2D6: *fluoxetine (Prozac®)

  * sertraline (Zoloft®)
  * paroxetine (Paxil®)
  * venlafaxine (Effexor®)
  * imipramine
  * nortriptyline
  * desipramine
  * amitriptyline
  * fenfluramine
  * terbinafine
  * cyclobenzaprine
  * haloperidol (Haldol®)
  * metoprolol
  * quinidine
  * propafenone (Rythmol®)
  * cimetidine (Tagamet®)
  * tamoxifen
  * over-the-counter diphenhydramine-containing drugs
  * including Benadryl and generics and the cough and cold preparations
  * Dytuss®
  * Tusstat®
  * Robitussin®
  * pro-drugs codeine
  * tramadol
  * hydrocodone
  * oxycodone (Percodan®, Percocet®) that are converted by 2D6 into their active forms.
* Illicit drug use, treatment within the past 2 months with paroxetine or fluoxetine, or the past six months with terbinafine are also exclusion criteria.
* Inability or unwillingness to fast 2 hours prior to the study session
* Existence of diagnosis which may influence absorption and gastric emptying; such as reflux , inflammatory bowel disease, or Crohn's disease.
* A demonstrated adverse reaction to previous dextromethorphan exposure
* Impaired hepatic or renal activity, or physical examination as determined by the Sub Investigator's discretion.
* Pregnancy
* Body-mass index (BMI) <5th percentile

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases: Pediatric patients who have a primary diagnosis of ADHD, combined type, hyperactive impulsive, or inattentive type (ADD). (110 subjects)
  Controls: Age and gender matched subjects who do not meet any of the exclusion criteria (110 subjects)
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Characterize the change in CYP2D6 and CYP3A4 phenotype through adolescence | Three years
  Growth and development adds an additional level of complexity as the genotype-phenotype relationship may change as children grow and develop. The purpose of this proposal is to characterize the relative roles of ontogeny and genetic variation towards changes in CYP2D6 and CYP3A4 activity during adolescence. Because some drugs commonly used to treat ADHD are metabolized by CYP2D6 and CYP3A4, the information gained from this study will contribute to a better understanding of the dosage requirements of medications used in this patient population.

SECONDARY OUTCOMES:
Identify endogenous markers of CYP2D6 activity | Three years
  Metabolomic strategies (HPLC-MS/MS) will be utilized to identify and characterize endogenous compounds that correlate with the formation of dextrorphan (CYP2D6 activity)from the parent compound, dextromethorphan, administered as a phenotyping probe.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Leeder, PharmD, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (2):
- United States (2):
  - The Children's Mercy Hospital, Kansas City, Missouri
  - The University of Washington, Seattle, Washington